CLINICAL TRIAL: NCT01296802
Title: Investigation of Serotonin Neurotransmission in "Ecstasy" Users Employing Combined Dexfenfluramine Challenge and Positron Emission Tomography: a Functional Probe to Assess MDMA Neurotoxicity
Brief Title: Investigation of Serotonin Neurotransmission in MDMA Users Using Combinated Dexfenfluramine Challenge and PET Imaging
Acronym: DEXFEN_PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Boris B. Quednow, Prof. Dr. Boris Quednow, University Hospital of Psychiatry Zurich., University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PUK_Study_72
Record Dates: First submitted 2011-02-07; First posted 2011-02-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Amphetamine-Related Disorders; Amphetamine Abuse
Keywords: Ecstasy; MDMA; Serotonin; Neurotoxicity; dexfenfluramine; Positron emission tomography; altanserin; 5-HT2A receptor
MeSH Terms: conditions — Amphetamine-Related Disorders; Neurotoxicity Syndromes | interventions — Dexfenfluramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: dexfenfluramine
- Dexfenfluramine (Experimental): Dexfenfluramine HCL
  Interventions: Drug: dexfenfluramine

INTERVENTIONS:
Drug: dexfenfluramine — oral, 40 mg to 60 mg, single application as a challenge
  Other Names: d-fenfluramine; Benzeneethanamine; (S)-N-Ethyl-1-[3-(trifluoromethyl)phenyl]-propan-2-amine

SUMMARY:
Illicit use of the psychostimulant "Ecstasy" (3,4-methylenedioxymethamphetamine, MDMA) is considered a major public health issue. In Switzerland, MDMA and congeners are - after cannabis and cocaine - number three in the ranking of the most popular illicit drugs. Worldwide, Ecstasy is estimated to be even the second most popular illicit drug, used by millions of regular users.

On the basis of animal data, it is likely that MDMA at high or cumulative doses damages serotonin (5-HT) neurons in the human brain. However, because of a multitude of methodological problems and a limited number of studies conducted in human subjects, no firm conclusions can yet be established whether chronic MDMA exposure produces a long lasting 5-HT deficiency syndrome, with consequent neuropsychiatric risks. To further address the putative neurotoxicity of MDMA in the human brain, we propose that novel functional assays of serotonergic neurotransmission may be useful to clarify this issue. We suggest that a 5-HT challenge study using positron emission tomography (PET) in conjunction with the 5-HT releaser dexfenfluramine [(+)FEN] may test the functional integrity of the 5-HT system in the living human brain.

Specifically, in a placebo-controlled study, the 5-HT release capacity of serotonergic neurons shall be investigated by assessing [18F]-altanserin binding to 5-HT2A receptors following (+)FEN challenge in former and continuing MDMA users, and age and sex-matched MDMA-naïve controls. (+)FEN is a potent serotonin releaser without relevant affinity for 5-HT, dopamine (DA) or norepinephrine (NE) receptors, and devoid of acute adverse effects in man. This makes (+)FEN an ideal pharmacological probe to explore functional integrity of serotonin neurotransmission.

A second aim of our investigation is to detect possible impairments of cognitive functions and to study their relationship to serotonin neurotransmission as indexed by PET. In the course of the neuroimaging study, the investigators therefore also measure cognitive (e.g. attention, visual and working memory, learning, executive function) and affective functions (e.g. anxiety, impulsivity), suspected to be altered due to chronic MDMA use. Using correlational analyses, the investigators aim to determine if circumscribed regions of altered 5-HT function are associated with specific impairments in cognitive and/or behavioural parameters.

We hypothesize that (+)FEN-evoked 5-HT release will discernibly alter availability of 5-HT2A receptors to [18F]-altanserin, with a pattern revealing the spatially heterogeneous vulnerability of 5-HT innervations to MDMA. The investigators predict that [18F]-altanserin volume of distribution (DV) will decline following (+)FEN challenge to a lesser extent in current MDMA users compared to MDMA-naïve control subjects. On the basis of animal data and recent neuroimaging studies in humans, the investigators hypothesize that functional recovery in former MDMA users will be manifest by a normalization or overshoot of the 5-HT release capacity.

Our methodology will allow us to quantitatively assess serotonergic functions in the living human brain. The novel combination of (+)FEN-induced release of 5-HT from intracellular storage vesicles and subsequent PET assessment of competitively altered [18F]-altanserin binding at postsynaptic 5-HT2A receptors will provide a more direct biological marker of in vivo serotonin function than has been hitherto available. By applying this new pharmacological challenge/PET neuroimaging approach to groups of current and former users of MDMA, the investigators shall be able to gain important new insight in the debated functional consequences of MDMA use, especially concerning the controversy about the reversibility of 5-HT changes following cessation of MDMA use. Successful completion of this project should have useful implications for public education and harm reduction with respect to MDMA use, and may also facilitate the development of possible treatment options for chronic MDMA users.

DETAILED DESCRIPTION:
Introduction: Illicit use of the psychostimulant 3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") is considered a major public health issue. In Switzerland, the proportion of teenage MDMA users has increased continuously in recent years. According to a representative survey from 2002, approximately 3.3% of the 15-16 year old students in Switzerland have taken MDMA at least once. Compared with the corresponding data from 1994 (1.8%) and 1998 (1.9%), the increase of MDMA use among is evident. In another survey from the Swiss Institute for the Prevention of Alcoholism and Drug Addiction (SFA/ISPA) 2.2% of the anonymously interviewed subjects between 15 to 39 years reported experiences with MDMA. Also worldwide, MDMA has become one of the most widely used illegal psychoactive drugs, with millions of regular users.

Acute administration of MDMA produces a rapid and marked release of serotonin (5-HT) via inhibition and reversal of the 5-HT transporter. Since the late 1980s, studies in non-human primates have provided convincing evidence that high doses of MDMA cause a substantial and sustained long-term neurotoxic loss of exclusively 5-HT nerve terminals with an associated depletion of up to 95% of 5-HT in several brain regions. In contrast, other neurotransmitter systems such as dopamine or norepinephrine remain undamaged. Subsequently, two studies with MDMA users have also shown selective decrements in cerebrospinal fluid (CSF) concentrations of 5-hydroxy indoleacetic acid, a marker for 5-HT depletion. In contrast, CSF concentrations of homovanillic acid or 3-methoxy-4-hydroxyphenylglycol, the major metabolites of dopamine and norepinephrine, were unchanged. Some imaging studies with serotonergic radioligands showed reduced 5-HT transporter (SERT) densities in cortical and subcortical brain regions of MDMA users. Moreover, electrophysiological studies have also suggested alterations of the 5-HT system in regular users of MDMA. However, most of these findings in humans have been strongly criticised for methodological flaws (e.g. small sample sizes or lack of specificity of the applied radioligands). Consequently, there is as yet no convincing evidence for a selective serotonergic neurotoxicity of MDMA in humans. Moreover, the mechanism of MDMA neurotoxicity in animals is still under debate.

In spite of these reservations, it has been consistently shown that MDMA users display dose-related impairments of verbal and visual-spatial memory, and impairments of executive functions and decision-making cognition. So far, the neuroanatomical basis of these neuropsychological deficits, and their relationship with 5-HT depletion, remain unclear.

On the basis of animal data, it is likely that MDMA at high or cumulative doses damages 5-HT neurons in the human brain. However, because of a multitude of methodological problems and a limited number of studies conducted in human subjects, no firm conclusions can yet be established whether chronic MDMA exposure produces a long lasting 5-HT deficiency syndrome, with consequent neuropsychiatric risks. To further address the putative neurotoxicity of MDMA in the human brain, we propose that, in addition to the present receptor mapping studies, novel functional assays of serotonergic neurotransmission may be useful to clarify this issue. Specifically, we suggest that 5-HT challenge studies using positron emission tomography (PET) in conjunction with the serotonin releaser dexfenfluramine [(+)FEN] may test the functional integrity of the 5-HT system in the living human brain.

Aims: To overcome impediments of previous imaging studies we propose to use a more direct approach to assess the integrity of serotonergic function in the human brain. 5-HT2A receptor mapping with PET and [18F]-altanserin, in combination with (+)FEN challenge, shall be used to investigate the 5-HT release capacity in current and former users of MDMA in comparison to drug-naïve control subjects.

We anticipate that the comparison of changed specific binding of [18F]-altanserin to 5-HT2A receptors following (+)FEN-induced 5-HT release will reveal whether chronic abuse of MDMA leads to functional alterations in the human brain, and if MDMA users face an increased risk of developing a chronic serotonin deficiency syndrome, possibly associated with cognitive impairment and depression or anxiety. Our biological marker for 5-HT function in vivo shall enable us to topographically map regional 5-HT release, and hence to determine if the hypothesized 5-HT depletion has global or focal consequences for the action of (+)FEN. The putative functional consequences (affect regulation, cognition, and behaviour) can be linked to regions of reduced 5-HT transmission.

By investigating current and former MDMA users, we shall assess the reversibility of 5-HT depletion. Furthermore, our (+)FEN challenge/PET imaging technique may reveal regions of increased 5-HT transmission due to hyperinnervation of 5-HT dendrites ("sprouting"), as occurs in MDMA-treated primates.

In the course of the PET study, we shall also measure cognitive (e.g. attention, visual and working memory, learning, executive function) and affective functions (e.g. anxiety, impulsivity), suspected to be altered due to chronic MDMA use. Using correlational analyses, we aim to determine if circumscribed regions of altered 5-HT function are associated with specific impairments in cognitive and/or behavioural parameters.

Current status of the project and pilot data: The radiosynthesis of the tracer [18F]-altanserin was established and validated according to GMP guidelines. The study and the use of (+)FEN and [18F]-altanserin has already been approved by the local ethics committee, Swissmedic and the Swiss Federal Office for Public Health (BAG). Furthermore, more than 50 present and former MDMA users and 20 drug-naïve control subjects have been screened, and found to meet general inclusion criteria. We applied our method to four healthy human volunteers to prove our concept. The PET scans were metabolite corrected and normalised according to Logans graphical method. The regions of interest-based analysis was done with PMOD. We found that the apparent distribution volume (DV) of [18F]-altanserin was strongly decreased in all brain regions by about 11 to 15%. Thus, the proposed method is suitable to investigate 5-HT release capacity in humans.

Working hypotheses: We hypothesize that (+)FEN-evoked 5-HT release will discernibly alter availability of 5-HT2A receptors to [18F]-altanserin, with a pattern revealing the spatially heterogeneous vulnerability of 5-HT innervations to MDMA. We predict that [18F]-altanserin DV will decline following (+)FEN challenge to a lesser extent in current MDMA users compared to MDMA-naïve control subjects. On the basis of animal data and recent neuroimaging studies in humans, we hypothesize that functional recovery in former MDMA users will be manifest by a normalization or overshoot of the serotonin release capacity.

5-HT neurotransmission will not be homogeneously reduced in chronic MDMA users, but that toxic effects will be most evident in the frontal cortex and subcortical structures such as caudate nucleus and thalamus; these regions are innervated by fine fibers arising from the dorsal raphe nuclei that are especially sensitive to MDMA neurotoxicity in non-human primates. Based on results of recent human studies, we furthermore anticipate a dose-related impairment of cognitive functions, especially of memory and learning, as well as an increased state anxiety in current MDMA users, followed by improvement after cessation of drug use, although recovery may be incomplete. Finally, we hypothesize that the degree of impairment of cognitive functions will correlate significantly with the measured reduction of 5-HT function.

Study design: To compare 5-HT neurotransmission in current MDMA users, former MDMA users, and MDMA-naïve control subjects, 16 subjects per group will be examined with [18F]-altanserin PET under two conditions. On two days - separated by an interval of 7 days - subjects will receive, in random order, placebo or 60 mg (+)FEN. Two hours later subjects will be positioned in the GE PET/CT with the head partially immobilized. Following acquisition of a low dose CT transmission scan, [18F]-altanserin (250 MBq, high specific activity) will be administered intravenously as a bolus over 30 sec, and dynamic PET data will be acquired during 90 minutes as a series of 36 frames increasing in duration from one minute to ten minutes. Subsequently, subjects will undergo a series of cognitive tasks from the Cambridge Neuropsychological Test Automated Battery (CANTAB). Moreover, potential affective reactions to the 5-HT release, anticipated group differences and the time course of affective reaction will be assessed by repeated use of psychometric questionnaires, specifically the State-Trait Anxiety Inventory (STAI), and Adjective Mood Rating Scale (AMRS). At intervals during the extended scanning and cognitive testing, venous blood samples will be collected for assay of (+)FEN, prolactin and cortisol concentrations by standard clinical procedures. The neuroendocrine responses will be correlated with the individual PET and neuropsychological test results.

Subjects and screening procedure: Participants for the study are recruited by means of flyers distributed at locations associated with the "techno" and "rave" scene in Zurich, with the help of local associations involved in drug prevention/information and harm reduction. Experimental groups are matched for sex, age, and cannabis use. Sixteen subjects of both genders, aged 18 to 35, will be recruited for each of the following three experimental groups: 1) Current MDMA users (self-estimated lifetime use of ≥ 50 tablets of "Ecstasy", the last intake is dated back within the last 4 weeks), 2) former MDMA users (self-estimated lifetime use of ≥ 50 tablets, but subjects will have stopped using Ecstasy for at least one year prior inclusion), and 3) MDMA-naïve control subjects.

Health of subjects will be determined by a general medical examination including electrocardiogram and standard laboratory parameters. To exclude subjects with current or past psychiatric conditions, all subjects will be assessed and diagnosed by a clinical psychologist using the SKID-I. During recruitments, potential subjects will be provided with extensive background information regarding administration of (+)FEN, neuropsychological testing, PET measures, and associated (radiation) risks, and will then be invited to give their written informed consent. Special liability is covered by hospital insurance for all subjects participating in this project. Pregnancy is an exclusion criterion; all female potential test subjects will have to agree to carry out a pregnancy test before entering the study.

A detailed history of psychoactive drug use, including type of drugs, first and last use, and estimated total use will be recorded. All subjects will have to agree to abstain from using any psychoactive drug (except nicotine and cannabis) for at least two weeks before the first PET scan. At the beginning of each of the two experimental days, urine samples will be collected and screened for the presence of psychoactive drugs or metabolites.

Relevance of the project: Our methodology will allow us to quantitatively assess serotonergic functions in the living human brain. The novel combination of (+)FEN-induced release of 5-HT from intracellular storage vesicles and subsequent PET assessment of competitively altered [18F]-altanserin binding at postsynaptic 5-HT2A receptors will provide a more direct biological marker of in vivo serotonin function than has been hitherto available. By applying this new pharmacological challenge/PET neuroimaging approach to groups of current and former users of MDMA, we shall be able to gain important new insight in the debated functional consequences of MDMA use, especially concerning the controversy about the reversibility of 5-HT changes following cessation of MDMA use. The topographic mapping of regional 5-HT release following (+)FEN challenge in two groups of MDMA users and in a drug-naïve cohort will help to assess the contentious issue if chronic MDMA users face the risk of developing a global 5-HT deficiency syndrome, characterized by cognitive and affective changes. Successful completion of this project should have useful implications for public education and harm reduction with respect to MDMA use, and may also facilitate the development of possible treatment options for chronic MDMA users.

ELIGIBILITY:
Inclusion Criteria:

* Current and former MDMA users: lifetime use of ≥ 50 tablets of Ecstasy
* Current MDMA users: Ecstasy use in the last 4 weeks
* Former MDMA users: at least 1 year of abstinence of Ecstasy and other psychostimulants
* MDMA-naïve control subjects: no lifetime use of MDMA or other psychostimulants

Exclusion Criteria:

* Female sex
* Positive drug urine screening (with exception for cannabis)
* Relevant somatic, neurological or psychiatric illness
* Current use of psychotropic medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Serotonin release capacity | 14 days
  [18F]-altanserin binding to 5-HT2A receptors following dexfenfluramine challenge compared to placebo

SECONDARY OUTCOMES:
Cognition | 14 day
  Changes in cognition (e.g., memory) after dexfenfluramine challenge compared to placebo
Prolactin and cortisol | 14 days
  Changes of prolactin and cortisol after dexfenfluramine challenge and placebo
Mood and mental state | 14 days
  Changes in mood and mental states after dexfenfluramine compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Franz X Vollenweider, Prof., Principal Investigator — University Hospital of Psychiatry Zurich; Boris B Quednow, Prof, Principal Investigator — University Hospital of Psychiatry Zurich
Locations (1):
- University Hospital of Psychiatry Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Hasler F, Kuznetsova OF, Krasikova RN, Cservenyak T, Quednow BB, Vollenweider FX, Ametamey SM, Westera G. GMP-compliant radiosynthesis of [18F]altanserin and human plasma metabolite studies. Appl Radiat Isot. 2009 Apr;67(4):598-601. doi: 10.1016/j.apradiso.2008.12.007. Epub 2008 Dec 24. PMID 19162492
- [Result] Quednow BB, Treyer V, Hasler F, Dorig N, Wyss MT, Burger C, Rentsch KM, Westera G, Schubiger PA, Buck A, Vollenweider FX. Assessment of serotonin release capacity in the human brain using dexfenfluramine challenge and [18F]altanserin positron emission tomography. Neuroimage. 2012 Feb 15;59(4):3922-32. doi: 10.1016/j.neuroimage.2011.09.045. Epub 2011 Oct 5. PMID 21996132